CLINICAL TRIAL: NCT06717945
Title: The Efficacy and Safety of Remimazolam Besylate for Cardiac Anesthesia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, director of department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No.2022-1786
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam besylate (Experimental): Patients received an initial dose of remimazolam (0.3mg/kg) for induction and a continuous infusion rate of 1 mg/kg/h for anesthesia maintenance.
  Interventions: Drug: remimazolam besylate
- propofol (Active Comparator): Patients received an initial dose of propofol (1.0 mg/kg) and a continuous infusion rate of 1-1.5 mg/kg/h
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: remimazolam besylate — Patients received an initial dose of remimazolam (0.3mg/kg) for induction and a continuous infusion rate of 1 mg/kg/h for anesthesia maintenance. Sedative was adjusted to maintain a bispectral index (BIS) at 40-60 after induction.
  Arms: remimazolam besylate
Drug: propofol — Patients received an initial dose of propofol (1.0 mg/kg) and a continuous infusion rate of 1-1.5 mg/kg/h. Sedative was adjusted to maintain a bispectral index (BIS) at 40-60 after induction.
  Arms: propofol

SUMMARY:
The evidence on the practice of remimazolam besylate during cardiac anesthesia is scarce. This study investigates the efficacy and safety of remimazolam besylate general induction and maintenance during cardiac surgery.

DETAILED DESCRIPTION:
Remimazolam besylate (RB), as a new benzodiazepine sedative agent, has been approved in clinical anesthesia with prominent characteristics of short onset/offset, less depression for cardiovascular or respiratory function and specific antagonist. Some studies have confirmed the comparable anesthesia efficacy of remimazolam for outpatient digestive endoscopy, fiberoptic bronchoscopy, facial plastic and orthopedic surgery as propofol. Currently, the evidence on its application in cardiac anesthesia is insufficient. Our study aims to evaluate the efficacy of remimazolam besylate and propofol and provide an ideal anesthetic agent to achieve the goal of early recovery after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective cardiac surgery via cardiopulmonary bypass;
2. Aged 18-65 years;
3. American Society of Anesthesiologists (ASA) grade I-III;
4. Body mass index (BMI) 18-28 kg/m2.

Exclusion Criteria:

1. A history of sternotomy for heart disease;
2. Angina or arrhythmia with severe dynamics flutters pre-operation;
3. Respiratory, hepatic or renal dysfunction (oxygenation index<300, alanine transaminase> 2 upper limits of normal value, creatinine > 200 μmol/L);
4. Diagnosed with advanced tumors;
5. Psychiatric or mental disorders;
6. Myasthenia gravis or seizures;
7. Pregnant or lactating females;
8. A history of benzodiazepines administration within 3 months before surgery;
9. Known allergic to benzodiazepines, opioids, propofol and flumazenil;
10. Involved in another interventional clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ratio of successful sedation during the whole surgery | Intraoperative period
  Sedation success is defined as BIS locating in the range of 40-60 according to the required dosage without additional rescue sedative during the surgical procedures.

SECONDARY OUTCOMES:
time interval for BIS from baseline before induction to 60 | Intraoperative period

IPD SHARING:
Plan to Share IPD: No